CLINICAL TRIAL: NCT02880163
Title: Reducing Exsanguination Via In-Vivo Expandable Foam
Brief Title: REVIVE: Reducing Exsanguination Via In-Vivo Expandable Foam
Acronym: REVIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arsenal Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-030
Record Dates: First submitted 2016-08-19; First posted 2016-08-26 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hemorrhagic Shock; Trauma; Exsanguinating Hemorrhage; Shock; Traumatic
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries; Exsanguination; Shock, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ResQFoam (Experimental): ResQFoam in-vivo expandable foam
  Interventions: Device: ResQFoam

INTERVENTIONS:
Device: ResQFoam — Hemostatic device for the treatment of emergent, exsanguinating, Class III or IV intraabdominal hemorrhagic shock in subjects due to trauma

SUMMARY:
The purpose of this study is to demonstrate safety, effectiveness and benefit-risk profile of ResQFoam for the inhospital treatment of exsanguinating, intraabdominal haemorrhage due to trauma in patients where emergent laparotomy is required.

ELIGIBILITY:
Inclusion Criteria:

1. Estimated age of 15 years or older (or subject weight estimated at greater than 50 kg if age is unknown)
2. Emergent, exsanguinating hemorrhage, from abdominal source as defined by:

   * Class III or IV hemorrhagic shock or
   * Assessment of Blood Consumption (ABC) score ≥ 2
3. Confirmation of abdominal hemorrhage by:

   * Direct visualization or
   * Positive Focused Assessment with Sonography in Trauma (FAST) or
   * Diagnostic Peritoneal Aspiration (DPA)
4. No other known, uncontrolled active sources of hemorrhage
5. Subject is intubated and sedated per local guidelines
6. Decision to administer foam is made within 30 minutes of admission to the emergency department.
7. Decision made to proceed to emergent laparotomy made within 30 minutes of admission to the emergency department.
8. Definitive surgical care is expected to occur within three hours of foam deployment
9. Subject must also be receiving concurrent transfusion of fluids or blood products.

   Exclusion Criteria:
10. Known or suspected major diaphragm injury
11. Known or suspected untreated pneumothorax
12. Known or suspected untreated hemothorax
13. Known or suspected blunt or penetrating cardiac or thoracic aortic trauma
14. Traumatic brain injury resulting in decapitation, visible brain matter or considered non- survivable based on initial physical exam
15. Received greater than five consecutive minutes of cardiopulmonary resuscitation in the pre-emergency department setting
16. Patients with Pulseless Electrical Activity
17. Known allergy to isocyanate
18. Known or suspected pregnancy
19. History of prior abdominal surgery or evidence of abdominal surgery (scars)
20. Disrupted abdominal wall that, in the opinion of the investigator would preclude ResQFoam from being adequately contained within the abdominal cavity
21. Subject in whom the abdominal aortic junctional tourniquet (AAJT) or Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) techniques have been used
22. Known Prisoners
23. Subjects with burns > 20% of total body surface area
24. Subject/legally authorized representative/subject family member purposefully opted out of participation in the study
25. Known Do Not Resuscitate order (DNR) or Physician Orders for Life Sustaining Treatment (POLST)
26. Known enrollment in another randomized, interventional study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure after deployment of ResQFoam over baseline value | All SBP assessments prior to deployment of IP through removal of IP and completion of laparotomy. Patient will be followed through hospital discharge or through Day 30, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Pritts, MD, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Maegele M. Effective approaches to address noncompressible torso hemorrhage. Curr Opin Crit Care. 2024 Jun 1;30(3):202-208. doi: 10.1097/MCC.0000000000001141. Epub 2024 Feb 28. PMID 38441108